CLINICAL TRIAL: NCT02807558
Title: A Biomarker-Directed Phase 2 Trial of SY-1425, a Selective Retinoic Acid Receptor Alpha Agonist, in Adult Patients With Acute Myeloid Leukemia (AML) or Myelodysplastic Syndrome (MDS)
Brief Title: A Biomarker-Directed Phase 2 Trial of Tamibarotene (SY-1425) in Participants With Acute Myeloid Leukemia or Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Syros Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SY-1425-201; 2017-000783-14 (EudraCT Number)
Record Dates: First submitted 2016-06-13; First posted 2016-06-21 (Estimated); Results first posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-11

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome
Keywords: AML; MDS; non-acute promyelocytic leukemia (non-APL); lower-risk myelodysplastic syndrome (LR-MDS)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — tamibarotene; Azacitidine; daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (6):
- R/R Non-APL AML or R/R HR-MDS: Tamibarotene Monotherapy (Experimental): Participants with R/R non-APL AML or R/R HR-MDS will receive tamibarotene at 6 mg/m^2/day in 2 divided doses on Days 1-28 of a 28-day cycle.
  Interventions: Drug: Tamibarotene
- Newly Diagnosed Non-APL AML: Tamibarotene Monotherapy (Experimental): Newly diagnosed, treatment-naive participants with non-APL AML who were unlikely to tolerate standard intensive chemotherapy will receive tamibarotene at 6 mg/m^2/day in 2 divided doses on Days 1-28 of a 28-day cycle.
  Interventions: Drug: Tamibarotene
- Newly Diagnosed Non-APL AML: Tamibarotene and Azacitidine (Experimental): Newly diagnosed, treatment-naive participants with non-APL AML who are unlikely to tolerate standard intensive chemotherapy will receive tamibarotene at 6 mg/m^2/day in 2 divided doses on Days 8-28 of a 28-day cycle, and azacitidine at 75 mg/m^2 once daily on Days 1-7 of a 28-day cycle.
  Interventions: Drug: Tamibarotene; Drug: Azacitidine
- LR-MDS: Tamibarotene Monotherapy (Experimental): Participants with transfusion-dependent LR-MDS without the del 5q abnormality who are refractory to erythropoietin (EPO) treatment or unlikely to respond to EPO treatment will receive tamibarotene at 6 mg/m^2/day in 2 divided doses on Days 1-28 of a 28-day cycle.
  Interventions: Drug: Tamibarotene
- R/R non-APL AML or R/R HR-MDS: Tamibarotene and Daratumumab (Experimental): Participants with R/R non-APL AML or R/R HR-MDS will receive tamibarotene at 6 mg/m^2/day in 2 divided doses during a 7-day lead-in and on Days 1-28 of a 28-day cycle. Participants will also receive daratumumab at 16 mg/kg starting on Cycle 1 Day 1 once weekly for 8 weeks, followed by dosing every 2 weeks for 16 weeks, followed by dosing every 4 weeks.
  Interventions: Drug: Tamibarotene; Drug: Daratumumab
- R/R non-APL AML: Tamibarotene and Azacitidine (Experimental): Participants with R/R non-APL AML will receive tamibarotene at 6 mg/m^2/day in 2 divided doses on Days 8-28 of a 28-day cycle, and azacitidine at 75 mg/m^2 once daily on Days 1-7 of a 28-day cycle.
  Interventions: Drug: Tamibarotene; Drug: Azacitidine

INTERVENTIONS:
Drug: Tamibarotene — Administered as oral tablets
  Other Names: SY-1425
Drug: Azacitidine — Administered via intravenous (IV) or subcutaneous (SC) infusion
  Other Names: Vidaza
  Arms: Newly Diagnosed Non-APL AML: Tamibarotene and Azacitidine; R/R non-APL AML: Tamibarotene and Azacitidine
Drug: Daratumumab — Administered via IV infusion
  Other Names: Darzalex
  Arms: R/R non-APL AML or R/R HR-MDS: Tamibarotene and Daratumumab

SUMMARY:
The purpose of this study is to determine the activity of tamibarotene in participants with relapsed/refractory (R/R) AML (administered as a monotherapy or in combination with azacitidine), R/R higher-risk MDS (HR-MDS) (administered as a monotherapy or in combination with daratumumab), newly diagnosed treatment naïve AML participants who are unlikely to tolerate standard intensive chemotherapy (administered as a monotherapy or in combination with azacitidine), or lower-risk MDS (LR-MDS) (administered as a monotherapy).

ELIGIBILITY:
Key Inclusion Criteria:

1. Must have:

   1. Relapsed and/or refractory non-APL AML that has failed to achieve a complete remission (CR) or partial remission (PR) following standard induction therapy, or has relapsed after any duration of CR or PR i. Must have measurable disease with bone marrow blasts ≥5%at screening
   2. Relapsed and/or refractory HR-MDS (High / Very High Risk, as defined by the Revised International Prognostic Scoring System (IPSS-R)) that has failed to achieve a CR or PR, or any hematologic improvement (HI, per IWG 2006 criteria) after standard therapy with hypomethylating agents (e.g., azacitidine, decitabine), or has relapsed after any duration of CR or PR or HI i. Must have measurable disease with bone marrow blasts >5% at screening
   3. Newly diagnosed, treatment-naïve non-APL AML in participants who, at the time of study entry are unlikely to tolerate standard intensive chemotherapy due to age, performance status, or comorbidities based on at least one of the following criteria:

      * i. Age ≥ 75 years old
      * ii. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 3
      * iii. Cardiac history of congestive heart failure (CHF) or documented ejection fraction (EF) ≤ 50%
      * iv. Pulmonary disease with diffusing capacity of lung for carbon monoxide ≤ 65% or Forced Expiratory Volume in 1 Second ≤ 65%
      * v. Creatinine clearance ≥ 30 milliliter (mL)/minute (min) to < 45 mL/min
      * vi. Hepatic impairment with total bilirubin > 1.5 to ≤ 3.0 x upper limit of normal (ULN)
      * vii. Any other comorbidity that the Investigator judges to be incompatible with intensive chemotherapy, and reviewed and approved by the Sponsor prior to enrollment
   4. Transfusion-dependent LR-MDS without the del 5q abnormality, in participants refractory to erythropoietin treatment or unlikely to respond to erythropoietin treatment (EPO >500).

      * i. LR-MDS: Very Low /Low / Intermediate Risk, as defined by IPSS-R.
      * ii.Red blood cell (RBC) transfusion-dependent anemia defined as no eight consecutive weeks without RBC transfusions within the 16 weeks prior to study entry, or ≥4 RBC transfusions within the 8 weeks prior to study entry.
      * iii.Refractory to or ineligible for erythropoiesis-stimulating agents (ESAs) is defined as RBC-Transfusion Dependence despite ESA treatment of ≥40,000 units/week recombinant human erythropoietin for 8 weeks or an equivalent dose of darbepoetin (150 µg/week) or serum EPO level >500 milliunits (mU)/mL in participants not previously treated with ESAs.
2. Participants must be evaluated for the RARA super-enhancer associated biomarker or RARA pathway associated biomarker at the time of study screening.

   a. Participants treated with tamibarotene monotherapy and in combination with daratumumab, and R/R AML participants treated with tamibarotene in combination with azacitidine must be positive as defined by a pre-determined cut-off
3. Must be amenable to serial bone marrow aspirates and peripheral blood sampling during the study.
4. ECOG Performance Status (PS) of 0, 1 or 2. For newly diagnosed AML participants < 75 years of age, ECOG 0-3; for ≥ 75 years of age, ECOG 0-2.
5. Adequate organ function as defined by:

   1. Total bilirubin ≤ 1.5 x the upper limit of normal (ULN), unless suspected to have Gilbert's disease. For newly diagnosed AML participants < 75 years of age, total bilirubin ≤ 3 x ULN; for ≥ 75 years of age, total bilirubin ≤ 1.5 x ULN.
   2. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN or ≤ 5 x ULN if documented liver infiltration with leukemia cells
   3. Serum creatinine ≤ 2.0 x ULN or calculated creatinine clearance ≥ 45 mL/min based on the Cockroft-Gault glomerular filtration rate estimation. For newly diagnosed AML participants < 75 years of age, creatinine clearance ≥ 30 mL/min; for ≥ 75 years of age, creatinine clearance ≥ 45 mL/min.
6. Discontinued use of chemotherapy, radiation therapy, or growth factors for at least 2 weeks prior to first study treatment, with the exception of hydroxyurea.
7. No investigational agents within 2 weeks prior to first study treatment.
8. No strong inducers of CYP3A4 within 2 weeks prior to first study treatment.
9. Resolved acute effects of any prior AML/MDS therapy to baseline or ≤ Grade 1 CTCAE severity.

Key Exclusion Criteria:

1. Acute promyelocytic leukemia (APL, M3 subtype of AML) or participants with a t(9:22) cytogenetic translocation.
2. Hyperleukocytosis (leukocytes ≥25 x 109/L) at study entry. The participants may be treated with hydroxyurea according to routine practice, and enroll in the study when the leukocyte count falls below 25 x 109/L.
3. Participants known to be refractory to platelet or packed red cell transfusions per Institutional Guidelines, or a participant who refuses blood product support.
4. Prior treatment with all-trans retinoic acid (ATRA) or systemic retinoid for the treatment of hematologic malignancy.
5. Tamibarotene and daratumumab combination only - Prior or concurrent exposure to daratumumab or other CD38 therapies.
6. Tamibarotene and daratumumab combination only - Participant has either of the following:

   1. Known chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) <50% of predicted normal. Note that FEV1 testing is required for participants suspected of having COPD and participants must be excluded if FEV1 is <50% of predicted normal.
   2. Known moderate or severe persistent asthma within the past 2 years, or uncontrolled asthma of any classification. Note that participants who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed to participate in the study.
7. Participants with active malignancy (not including basal cell carcinoma, non-melanoma skin cancer, cervical carcinoma in situ, localized prostate cancer treated with hormone therapy). Participants with history of other cancers should be free of disease for at least 2 years.
8. Participants with hypertriglyceridemia defined as >1000 mg/dL (CTCAE Grade 4).
9. Participants with clinically significant cardiac disease including one of the following currently or in the previous 6 months: myocardial infarction, unstable cardiac function due to unstable angina or congestive heart failure, congenital long QT syndrome, torsades de pointes or significant ventricular arrhythmias.
10. Participants with known active uncontrolled central nervous system (CNS) leukemia.
11. Participants taking Vitamin A supplements (>10,000 IU/d) unless discontinued prior to first dose of study drug, or having hypervitaminosis.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Syros Pharmaceuticals
Locations (26):
- United States (14):
  - Hartford, Connecticut
  - Miami, Florida
  - Iowa City, Iowa
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - New York, New York
  - Rochester, New York
  - Durham, North Carolina
  - Cleveland, Ohio
  - Portland, Oregon
  - Allentown, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Nashville, Tennessee
  - Houston, Texas
- France (12):
  - CHU Amiens, Amiens
  - Centre Hospitalier de la Côte basque, Bayonne
  - Centre Hospitalier Universitiaire Hopital Avicenne, Bobigny
  - Hospital Morvan, Brest
  - Centre Hospitalier de Versailles - Hôpital André Mignot, Le Chesnay
  - Centre hospitalier Lyon Sud, Lyon
  - Centre Hospitalier Universitaire Nantes, Nantes
  - Nice Hospital, Archet Hospital 1 Clinical Hematology Service, Nice
  - Hopital Saint Louis, Paris
  - Hôpital Haut Leveque, Centre Francois Magendie, Pessac
  - Centre Hospitalier Universitaire Nancy, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Botton S, Cluzeau T, Vigil C, Cook RJ, Rousselot P, Rizzieri DA, Liesveld JL, Fenaux P, Braun T, Banos A, Jurcic JG, Sekeres MA, Savona MR, Roboz GJ, Bixby D, Madigan K, Volkert A, Stephens K, Kang-Fortner Q, Baker K, Paul S, McKeown M, Carulli J, Eaton M, Hodgson G, Fiore C, Kelly MJ, Roth DA, Stein EM. Targeting RARA overexpression with tamibarotene, a potent and selective RARalpha agonist, is a novel approach in AML. Blood Adv. 2023 May 9;7(9):1858-1870. doi: 10.1182/bloodadvances.2022008806. PMID 36477975

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Screening assessments were conducted within 30 days of dosing.
Groups:
- R/R Non-APL AML or R/R HR-MDS: Tamibarotene Monotherapy: Participants with Relapsed/Refractory (R/R) Non-Acute Promyelocytic Leukemia (APL) Acute Myeloid Leukemia (AML) or R/R Higher-risk Myelodysplastic Syndrome (HR-MDS) received tamibarotene at 6 milligrams (mg)/meter (m)^2/day in 2 divided doses on Days 1-28 of a 28-day cycle.
- Newly Diagnosed Non-APL AML: Tamibarotene Monotherapy: Newly diagnosed, treatment-naive participants with non-APL AML who were unlikely to tolerate standard intensive chemotherapy received tamibarotene at 6 mg/m^2/day in 2 divided doses on Days 1-28 of a 28- day cycle.
- LR-MDS: Tamibarotene Monotherapy: Participants with transfusion-dependent lower-risk myelodysplastic syndrome (LR-MDS) without the del- 5q abnormality who were refractory to erythropoietin (EPO) treatment or unlikely to respond to EPO treatment received tamibarotene at 6 mg/m^2/day in 2 divided doses from Days 1-28 of a 28-day cycle.
- Newly Diagnosed Non-APL AML: Tamibarotene and Azacitidine: Newly diagnosed, treatment-naive participants with non-APL AML who were unlikely to tolerate standard intensive chemotherapy received tamibarotene at 6 mg/m^2/day in 2 divided doses on Days 8-28 of a 28-day cycle, and azacitidine at 75 mg/m^2 once daily on Days 1-7 of a 28-day cycle.
- R/R Non-APL AML: Tamibarotene and Azacitidine: Participants with R/R non-APL AML received tamibarotene at 6 mg/m^2/day in 2 divided doses on Days 8-28 of a 28-day cycle, and azacitidine at 75 mg/m^2 once daily on Days 1-7 of a 28-day cycle.
- R/R Non-APL AML or R/R HR-MDS: Tamibarotene and Daratumumab: Participants with R/R non-APL AML or R/R HR-MDS received tamibarotene at 6 mg/m^2/day in 2 divided doses during a 7-day lead-in and on Days 1-28 of a 28-day cycle. Participants also received daratumumab at 16 mg/kg starting on Cycle 1 Day 1 once weekly for 8 weeks, followed by dosing every 2 weeks for 16 weeks, followed by dosing every 4 weeks.
Period: Overall Study
Arm/Group | R/R Non-APL AML or R/R HR-MDS: Tamibarotene Monotherapy | Newly Diagnosed Non-APL AML: Tamibarotene Monotherapy | LR-MDS: Tamibarotene Monotherapy | Newly Diagnosed Non-APL AML: Tamibarotene and Azacitidine | R/R Non-APL AML: Tamibarotene and Azacitidine | R/R Non-APL AML or R/R HR-MDS: Tamibarotene and Daratumumab
Started | 29 | 2 | 29 | 51 | 28 | 16
Received at Least 1 Dose of Study Drug | 29 | 2 | 29 | 51 | 28 | 16
Response Evaluable Population | 22 | 2 | 27 | 46 | 21 | 12
Completed Per Study Protocol | 29 | 2 | 29 | 51 | 27 | 16
Completed Post-Treatment Follow-up | 1 | 0 | 0 | 6 | 1 | 0
Evaluable for Hematological Improvement (HI) | 16 | 2 | 25 | 16 | 17 | 9
Completed | 1 | 0 | 0 | 6 | 2 | 0
Not Completed | 28 | 2 | 29 | 45 | 26 | 16
Not completed — Consent withdrawn by participant | 4 | 0 | 4 | 2 | 1 | 0
Not completed — Non-compliance with Study Drug | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 9 | 0 | 0 | 0
Not completed — Death | 23 | 2 | 3 | 43 | 24 | 15
Not completed — Progressive Disease | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Other than specified | 1 | 0 | 2 | 0 | 1 | 1
Not completed — Lack of Efficacy | 0 | 0 | 9 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all screened participants who received any amount of study drug (tamibarotene or combination treatment).
Groups:
- R/R Non-APL AML or R/R HR-MDS: Tamibarotene Monotherapy: Participants with R/R non-APL AML or R/R HR-MDS received tamibarotene at 6 mg/m^2/day in 2 divided doses on Days 1-28 of a 28-day cycle.
- LR-MDS: Tamibarotene Monotherapy: Participants with transfusion-dependent LR-MDS without the del- 5q abnormality who were refractory to EPO treatment or unlikely to respond to EPO treatment received tamibarotene at 6 mg/m^2/day in 2 divided doses from Days 1-28 of a 28-day cycle.
- Total: Total of all reporting groups
Arm/Group | R/R Non-APL AML or R/R HR-MDS: Tamibarotene Monotherapy | Newly Diagnosed Non-APL AML: Tamibarotene Monotherapy | LR-MDS: Tamibarotene Monotherapy | Newly Diagnosed Non-APL AML: Tamibarotene and Azacitidine | R/R Non-APL AML: Tamibarotene and Azacitidine | R/R Non-APL AML or R/R HR-MDS: Tamibarotene and Daratumumab | Total
Number analyzed (Participants) | 29 | 2 | 29 | 51 | 28 | 16 | 155
Age, Customized [Count of Participants; unit: Participants]
  Adults (18-64 years) | 5 | 0 | 2 | 3 | 5 | 5 | 20
  From 65-84 years | 21 | 2 | 24 | 43 | 21 | 11 | 122
  85 years and over | 3 | 0 | 3 | 5 | 2 | 0 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 0 | 10 | 19 | 15 | 8 | 64
  Male | 17 | 2 | 19 | 32 | 13 | 8 | 91
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 2 | 6 | 3 | 2 | 18
  Not Hispanic or Latino | 25 | 0 | 25 | 29 | 16 | 13 | 108
  Unknown or Not Reported | 1 | 0 | 2 | 16 | 9 | 1 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 2 | 1 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 3 | 2 | 0 | 0 | 8
  White | 25 | 0 | 22 | 30 | 18 | 14 | 109
  More than one race | 0 | 1 | 1 | 2 | 0 | 0 | 4
  Unknown or Not Reported | 0 | 1 | 3 | 15 | 9 | 2 | 30

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) in Biomarker Positive AML or HR-MDS Participants Treated With Tamibarotene Monotherapy or in Combination With Azacitidine
Description: ORR was defined as: AML: number of participants with complete remission (CR), CR with incomplete blood count recovery (CRi), CR with partial hematologic recovery (CRh), partial remission(PR), or morphologic leukemia-free state (MLFS) determined by the investigator per revised International Working Group (IWG) AML criteria. HR-MDS: the number of participants with CR, PR, marrow CR (mCR), or HI determined by the investigator per revised IWG MDS criteria.
Time Frame: Up to 48 months
Population: Response Evaluable Population included participants who completed 1 cycle of study treatment, and had a follow-up assessment of disease status, and did not have any major protocol violations, or withdrew from the study before completion of Cycle 1 because of documented disease progression. Overall Number of Participants analyzed (N) = participants evaluable for this Outcome Measure.
Measure: Count of Participants; unit: Participants
Groups:
- ND Non-APL AML: Tamibarotene and Azacitidine: RARA-Positive: Participants from the "Newly Diagnosed Non-APL AML: Tamibarotene and Azacitidine" arm who were positive for the retinoic acid receptor alpha (RARA) super-enhancer associated biomarker (RARA-positive) were included in this subgroup analysis.
  Participants who were unlikely to tolerate standard intensive chemotherapy received tamibarotene at 6 mg/m^2/day in 2 divided doses on Days 8-28 of a 28-day cycle, and azacitidine at 75 mg/m^2 once daily on Days 1-7 of a 28-day cycle.
Arm/Group | R/R Non-APL AML or R/R HR-MDS: Tamibarotene Monotherapy | Newly Diagnosed Non-APL AML: Tamibarotene Monotherapy | R/R Non-APL AML: Tamibarotene and Azacitidine | ND Non-APL AML: Tamibarotene and Azacitidine: RARA-Positive
Number analyzed (Participants) | 22 | 2 | 21 | 18
Participants | 2 | 0 | 4 | 12

2. Primary Outcome: Transfusion Independence Rate (TIR) for LR-MDS Participants Treated With Tamibarotene Monotherapy
Description: TIR was defined as the number of participants who achieved transfusion independence defined as 8 consecutive weeks of red blood cell (RBC) transfusion independence.
Time Frame: Up to 48 months
Population: Population evaluable for TIR, which included all participants who received at least 8 weeks of study treatment.
  Here, Overall Number of Participants analyzed (N) = participants evaluable for this Outcome Measure.
Measure: Count of Participants; unit: Participants
Groups:
- LR-MDS: Tamibarotene Monotherapy: Participants with transfusion-dependent LR-MDS without the del-5q abnormality who were refractory to EPO treatment or unlikely to respond to EPO treatment received tamibarotene at 6 mg/m^2/day in 2 divided doses from Days 1-28 of a 28-day cycle.
Arm/Group | LR-MDS: Tamibarotene Monotherapy
Number analyzed (Participants) | 27
Participants | 0

3. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) Treated With Tamibarotene in Combination With Daratumumab
Description: A TEAE was any untoward medical occurrence associated with use of a study drug/study participation, whether or not considered related to study drug after first dose. A TEAE was any unfavorable/unintended sign (including abnormal laboratory finding), symptom, or disease temporally associated with the study drug. A serious TEAE resulted in death, was life-threatening, required inpatient hospitalization/prolongation of existing hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect in the offspring of a participant who received study drug or other important medical events. A summary of serious and all other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Up to 48 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | R/R Non-APL AML or R/R HR-MDS: Tamibarotene and Daratumumab
Number analyzed (Participants) | 16
Participants
  TEAE | 16
  Treatment-emergent Serious Adverse Event (SAE) | 12

4. Secondary Outcome: ORR in AML Participants Positive for the RARA Super-enhancer Associated Biomarker Treated With Tamibarotene in Combination With Azacitidine
Description: ORR was defined as: AML: the number of participants with CR, CRi, CRh, PR, or MLFS as determined by the investigator per the revised IWG AML criteria.
  Per prespecified analysis, data were not collected for this Outcome Measure for the "R/R Non-APL AML or R/R HR-MDS: Tamibarotene Monotherapy" arm, the "Newly Diagnosed Non-APL AML: Tamibarotene Monotherapy" arm, and the "R/R non-APL AML or R/R HR-MDS: Tamibarotene and Daratumumab" arm as there were fewer than 5 responders per arm. Data are presented per specifications in the statistical analysis plan.
Time Frame: Up to 48 months
Population: Response evaluable population (which included participants who completed 1 cycle of study treatment, and had a follow-up assessment of disease status, and did not have any major protocol violations, or withdrew from the study before completion of Cycle 1 because of documented disease progression) in participants who were RARA-positive. Overall Number of Participants analyzed (N) = participants evaluable for this Outcome Measure.
Measure: Count of Participants; unit: Participants
Groups:
- ND Non-APL AML: Tamibarotene and Azacitidine: RARA-Positive: Participants from the "Newly Diagnosed Non-APL AML: Tamibarotene and Azacitidine" arm who were positive for the RARA super-enhancer associated biomarker (RARA-positive) were included in this subgroup analysis.
  Participants who were unlikely to tolerate standard intensive chemotherapy received tamibarotene at 6 mg/m^2/day in 2 divided doses on Days 8-28 of a 28-day cycle, and azacitidine at 75 mg/m^2 once daily on Days 1-7 of a 28-day cycle.
Arm/Group | R/R Non-APL AML: Tamibarotene and Azacitidine | ND Non-APL AML: Tamibarotene and Azacitidine: RARA-Positive
Number analyzed (Participants) | 21 | 18
Participants | 4 | 12

5. Secondary Outcome: ORR in AML Participants Positive for the Interferon Regulatory Factor 8 (IRF8) Biomarker and Negative for the RARA Super-enhancer Associated Biomarker Treated With Tamibarotene in Combination With Azacitidine
Description: ORR was defined as: AML: number of participants with CR, CRi, CRh, PR, or MLFS determined by the investigator per the revised IWG AML criteria.
  Per prespecified analysis, data were collected for this Outcome Measure only for the arm that enrolled the IRF8-positive participants and that included 5 or more responders. Data are presented per specifications in the statistical analysis plan.
Time Frame: Up to 48 months
Population: Response Evaluable Population (which included participants who completed 1 cycle of study treatment, had a follow-up assessment of disease status, did not have any major protocol violations or withdrew from study before completion of Cycle 1 because of documented disease progression) in participants who were positive for the IRF8 biomarker and negative for the RARA superenhancer associated biomarker. Overall Number of Participants analyzed (N) = participants evaluable for this Outcome Measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Newly Diagnosed Non-APL AML: Tamibarotene and Azacitidine
Number analyzed (Participants) | 4
Participants | 2

6. Secondary Outcome: ORR in AML Participants Negative for the RARA Super-enhancer Associated Biomarker Treated With Tamibarotene in Combination With Azacitidine
Description: ORR was defined as:
  AML: the number of participants with CR, CRi, CRh, PR, or MLFS as determined by the investigator per the revised IWG AML criteria.
  Per prespecified analysis, data were collected for this Outcome Measure only for the arm that enrolled the RARA-negative participants and that included 5 or more responders. Data are presented per specifications in the statistical analysis plan.
Time Frame: Up to 48 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- ND Non-APL AML: Tamibarotene and Azacitidine: RARA-Negative: Participants from the "Newly Diagnosed Non-APL AML:Tamibarotene and Azacitidine" arm who were negative for the RARA super-enhancer associated biomarker (RARA-negative) were included in this subgroup analysis.
  Participants who were unlikely to tolerate standard intensive chemotherapy received tamibarotene at 6 mg/m^2/day in 2 divided doses on Days 8-28 of a 28-day cycle, and azacitidine at 75 mg/m^2 once daily on Days 1-7 of a 28-day cycle.
Arm/Group | ND Non-APL AML: Tamibarotene and Azacitidine: RARA-Negative
Number analyzed (Participants) | 28
Participants | 12

7. Secondary Outcome: ORR for AML or HR-MDS Participants Treated With Tamibarotene in Combination With Daratumumab
Description: ORR was defined as:
  AML: the number of participants with CR, CRi, CRh, PR, or MLFS as determined by the investigator per the revised IWG AML criteria.
  HR-MDS: the number of participants with CR, PR, mCR, or HI as determined by the investigator per the revised IWG MDS criteria.
Time Frame: Up to 48 months
Population: Response evaluable population (which included participants who completed 1 cycle of study treatment, and had a follow-up assessment of disease status, and did not have any major protocol violations, or withdrew from the study before completion of Cycle 1 because of documented disease progression) who had evaluable data for the Outcome Measure.
Measure: Count of Participants; unit: Participants
Arm/Group | R/R Non-APL AML or R/R HR-MDS: Tamibarotene and Daratumumab
Number analyzed (Participants) | 12
Participants | 2

8. Secondary Outcome: Event-Free Survival (EFS) in AML and HR-MDS Participants Treated With Tamibarotene Monotherapy, or in Combination With Azacitidine or Daratumumab
Description: EFS was defined as time from first treatment until date of documentation of disease relapse following CR, CRi, or death, whichever occurred first. If the participant did not achieve a CR, EFS was defined as the point of progression or death, whichever occurred first.
  Per prespecified analysis, data were not collected for the Newly Diagnosed Non-APL AML: Tamibarotene Monotherapy arm as there were fewer than 5 participants in the arm. Additionally, per prespecified analysis, data were not collected for this Outcome Measure for the LR-MDS: Tamibarotene Monotherapy arm.
  Data are presented per specifications in the statistical analysis plan. All-cause mortality is reported in the Reported Adverse Events module.
Time Frame: Up to 48 months
Population: Safety population included all screened participants who received any amount of study drug (tamibarotene or combination treatment). Overall Number of Participants analyzed (N) = participants evaluable for this Outcome Measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | R/R Non-APL AML or R/R HR-MDS: Tamibarotene Monotherapy | R/R Non-APL AML: Tamibarotene and Azacitidine | R/R Non-APL AML or R/R HR-MDS: Tamibarotene and Daratumumab | ND Non-APL AML: Tamibarotene and Azacitidine: RARA-Positive | ND Non-APL AML: Tamibarotene and Azacitidine: RARA-Negative
Number analyzed (Participants) | 29 | 28 | 16 | 22 | 29
months | 2.6 [1.2 to 2.8] | 3.3 [1.9 to 5.5] | 1.2 [1.1 to 2.1] | 8.3 [3.1 to 11.8] | 6.6 [2.4 to 9.1]

9. Secondary Outcome: Duration of Response (DOR) in AML Participants Treated With Tamibarotene in Combination With Azacitidine
Description: DOR was defined as time from first date of response CR, CRi, CRh, MLFS or PR until the date of relapse.
  As prespecified, data were not collected for this Outcome Measure for any of the Tamibarotene Monotherapy arms, or R/R non-APL AML or R/R HR-MDS: Tamibarotene and Daratumumab arm.
  Data is presented as specified in the statistical analysis plan.
Time Frame: Up to 48 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | R/R Non-APL AML: Tamibarotene and Azacitidine | ND Non-APL AML: Tamibarotene and Azacitidine: RARA-Positive | ND Non-APL AML: Tamibarotene and Azacitidine: RARA-Negative
Number analyzed (Participants) | 21 | 18 | 28
months | 5.9 [1.0 to NA] — Upper confidence interval was not estimable by Brookmeyer and Crowley method due to insufficient observed events. | 10.8 [2.9 to NA] — Upper confidence interval was not estimable by Brookmeyer and Crowley method due to insufficient observed events. | 4.7 [2.5 to 32.3]

10. Secondary Outcome: Overall Survival (OS) in AML and HR-MDS Participants Treated With Tamibarotene Monotherapy, or in Combination With Azacitidine or Daratumumab
Description: OS was defined as the time from first treatment until death from any cause.
  Per planned analysis, data were not collected for this Outcome Measure for the Newly Diagnosed Non-APL AML: Tamibarotene Monotherapy arm as there were fewer than 5 participants in the study arm. Additionally, per prespecified analysis, data were not collected for this Outcome Measure for the LR-MDS: Tamibarotene Monotherapy arm.
  Data is presented as specified in the statistical analysis plan. All-cause mortality is reported in the Reported Adverse Events module.
Time Frame: Up to 48 months
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | R/R Non-APL AML or R/R HR-MDS: Tamibarotene Monotherapy | R/R Non-APL AML: Tamibarotene and Azacitidine | R/R Non-APL AML or R/R HR-MDS: Tamibarotene and Daratumumab | ND Non-APL AML: Tamibarotene and Azacitidine: RARA-Positive | ND Non-APL AML: Tamibarotene and Azacitidine: RARA-Negative
Number analyzed (Participants) | 29 | 28 | 16 | 22 | 29
months | 5.7 [2.7 to 7.1] | 5.9 [2.7 to 11.0] | 3.6 [1.8 to 4.6] | 8.4 [5.2 to 15.6] | 11.7 [6.6 to 15.8]

11. Secondary Outcome: Hematologic Improvement (HI) in AML, HR-MDS and LR-MDS Participants Treated With Tamibarotene Monotherapy, or in Combination With Azacitidine or Daratumumab
Description: HI was defined according to the modified IWG response criteria for MDS as the number of participants with a response (lasting at least 8 weeks) after first treatment, including erythroid response, platelet response, or neutrophil response.
  Data are presented per specifications in the statistical analysis plan.
Time Frame: Up to 48 months
Population: Measured in the population evaluable for HI, which included all participants who received at least 8 weeks of study treatment.
  Overall Number of Participants analyzed (N) = participants evaluable for this Outcome Measure.
Measure: Count of Participants; unit: Participants
Groups:
- ND Non-APL AML: Tamibarotene and Azacitidine: RARA-Negative: Participants from the "Newly Diagnosed Non-APL AML: Tamibarotene and Azacitidine" arm who were positive for the RARA super-enhancer associated biomarker (RARA-positive) were included in this subgroup analysis.
  Participants who were unlikely to tolerate standard intensive chemotherapy received tamibarotene at 6 mg/m^2/day in 2 divided doses on Days 8-28 of a 28-day cycle, and azacitidine at 75 mg/m^2 once daily on Days 1-7 of a 28-day cycle.
Arm/Group | R/R Non-APL AML or R/R HR-MDS: Tamibarotene Monotherapy | Newly Diagnosed Non-APL AML: Tamibarotene Monotherapy | LR-MDS: Tamibarotene Monotherapy | R/R Non-APL AML: Tamibarotene and Azacitidine | R/R Non-APL AML or R/R HR-MDS: Tamibarotene and Daratumumab | ND Non-APL AML: Tamibarotene and Azacitidine: RARA-Positive | ND Non-APL AML: Tamibarotene and Azacitidine: RARA-Negative
Number analyzed (Participants) | 16 | 2 | 25 | 17 | 9 | 16 | 19
Participants | 3 | 0 | 1 | 1 | 0 | 4 | 3

12. Secondary Outcome: Number of Participants With TEAEs in AML and MDS Participants Treated With Tamibarotene Monotherapy or in Combination With Azacitidine
Description: as for outcome 3
Time Frame: Up to 48 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | R/R Non-APL AML or R/R HR-MDS: Tamibarotene Monotherapy | Newly Diagnosed Non-APL AML: Tamibarotene Monotherapy | LR-MDS: Tamibarotene Monotherapy | Newly Diagnosed Non-APL AML: Tamibarotene and Azacitidine | R/R Non-APL AML: Tamibarotene and Azacitidine
Number analyzed (Participants) | 29 | 2 | 29 | 51 | 28
Participants
  TEAE | 29 | 2 | 29 | 51 | 27
  Treatment-emergent SAE | 16 | 2 | 15 | 43 | 20

ADVERSE EVENTS:
Time Frame: Up to 48 months
Description: Safety population included all screened participants who received any amount of study drug (tamibarotene or combination treatment).
Arm/Group | R/R Non-APL AML or R/R HR-MDS: Tamibarotene Monotherapy | Newly Diagnosed Non-APL AML: Tamibarotene Monotherapy | LR-MDS: Tamibarotene Monotherapy | Newly Diagnosed Non-APL AML: Tamibarotene and Azacitidine | R/R Non-APL AML: Tamibarotene and Azacitidine | R/R Non-APL AML or R/R HR-MDS: Tamibarotene and Daratumumab
All-Cause Mortality (participants affected / at risk) | 23/29 | 2/2 | 3/29 | 43/51 | 24/28 | 15/16
Serious Adverse Events (participants affected / at risk) | 16/29 | 2/2 | 15/29 | 43/51 | 20/28 | 12/16
Other Adverse Events (participants affected / at risk) | 29/29 | 2/2 | 29/29 | 50/51 | 27/28 | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | R/R Non-APL AML or R/R HR-MDS: Tamibarotene Monotherapy (N=29) | Newly Diagnosed Non-APL AML: Tamibarotene Monotherapy (N=2) | LR-MDS: Tamibarotene Monotherapy (N=29) | Newly Diagnosed Non-APL AML: Tamibarotene and Azacitidine (N=51) | R/R Non-APL AML: Tamibarotene and Azacitidine (N=28) | R/R Non-APL AML or R/R HR-MDS: Tamibarotene and Daratumumab (N=16)
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 2 | 0 | 0
Vasculitis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 5 | 1 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 0 | 0
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 3 | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 0
Cranial nerve disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Lacunar stroke (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Partial seizures (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | 0 | 0 | 12 | 9 | 7
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Leukostasis syndrome (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neutropenic colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Renal injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0 | 2 | 1 | 1
Pharyngeal abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 4 | 8 | 3 | 3
Pneumonia fungal (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 0
Pneumonia parainfluenzae viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pseudomonal sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 2 | 0 | 3 | 5 | 4 | 3
Septic shock (Infections and infestations) | 1 | 0 | 1 | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 1 | 1 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Klebsiella bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pseudomonas infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary mycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Arthritis infective (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Enterobacter pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Lung abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Malaria (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Nocardiosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Proteus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Serratia sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Streptococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cardiac Failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | R/R Non-APL AML or R/R HR-MDS: Tamibarotene Monotherapy (N=29) | Newly Diagnosed Non-APL AML: Tamibarotene Monotherapy (N=2) | LR-MDS: Tamibarotene Monotherapy (N=29) | Newly Diagnosed Non-APL AML: Tamibarotene and Azacitidine (N=51) | R/R Non-APL AML: Tamibarotene and Azacitidine (N=28) | R/R Non-APL AML or R/R HR-MDS: Tamibarotene and Daratumumab (N=16)
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Superficial spreading melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Pallor (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vascular insufficiency (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 0
Venous thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 3 | 0 | 1
Hypotension (Vascular disorders) | 2 | 0 | 2 | 6 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 3 | 2 | 0 | 0
Haematoma (Vascular disorders) | 0 | 2 | 0 | 0 | 4 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Erythema (Vascular disorders) | 1 | 0 | 2 | 1 | 0 | 0
Shoulder arthroplasty (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0
Adverse drug reaction (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 4 | 0 | 1 | 11 | 5 | 0
Catheter site erythema (General disorders) | 1 | 0 | 0 | 0 | 0 | 1
Catheter site pain (General disorders) | 1 | 0 | 0 | 1 | 0 | 1
Chills (General disorders) | 4 | 0 | 1 | 2 | 4 | 0
Crepitations (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Device related thrombosis (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Exercise tolerance decreased (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 2 | 0 | 0 | 0
Fatigue (General disorders) | 12 | 0 | 9 | 19 | 9 | 4
Gait disturbance (General disorders) | 0 | 1 | 1 | 1 | 0 | 1
Injection site bruising (General disorders) | 1 | 0 | 1 | 0 | 0 | 0
Injection site haemorrhage (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 1 | 0 | 3 | 2 | 0 | 0
Medical device pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Medical device site erythema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 8 | 1 | 5 | 19 | 4 | 4
Pain (General disorders) | 2 | 0 | 2 | 2 | 0 | 1
Pyrexia (General disorders) | 8 | 0 | 3 | 17 | 6 | 1
Catheter site rash (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 1 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Impaired healing (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Inflammatory pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 3 | 0 | 0
Injection site irritation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Injection site nodule (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 1 | 3 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 2 | 1 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 2 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 2 | 2 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 0 | 1 | 1 | 0
Catheter site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Early satiety (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Acute graft versus host disease (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vulvovaginal pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ovarian vein thrombosis (Reproductive system and breast disorders) | 0 | 0 | 1 | 1 | 0 | 0
Perineal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 1 | 4 | 9 | 3 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 0 | 2 | 13 | 6 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 2 | 5 | 7 | 2
Hypopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 1 | 2 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 2 | 3 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 4 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 2 | 3 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 3 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 2 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 2 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 1
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Acute promyelocytic leukaemia differentiation syndrome (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nasal mucosal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 6 | 2 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 2 | 4 | 0 | 0
Delirium (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 3 | 0
Depression (Psychiatric disorders) | 1 | 0 | 3 | 4 | 0 | 2
Hallucination (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 1 | 6 | 2 | 2
Hallucination, Visual acuity reduced (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Psychomotor retardation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 0
Genito-pelvic pain/penetration disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hallucination, Olfactory (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 3 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1 | 4 | 2 | 1
Amylase increased (Investigations) | 2 | 1 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 2 | 2 | 2 | 1
Blood cholesterol increased (Investigations) | 1 | 0 | 1 | 1 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 3 | 4 | 2 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Breath sounds abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Cardiac murmur (Investigations) | 2 | 0 | 0 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
High density lipoprotein decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 3 | 0 | 0 | 2
Lipase decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 2 | 0 | 2 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 4 | 1 | 0 | 1
Platelet count decreased (Investigations) | 3 | 0 | 1 | 4 | 0 | 1
Respiratory rate increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Skin turgor decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Vitamin K decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 6 | 1 | 6 | 18 | 5 | 1
White blood cell count decreased (Investigations) | 1 | 0 | 3 | 2 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 2 | 2 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Coronavirus test positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Respiratory syncytial virus test positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Troponin I increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 2 | 0 | 5 | 2 | 0 | 1
Chest X-ray abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Heart rate irregular (Investigations) | 0 | 0 | 0 | 0 | 0 | 2
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 3 | 0 | 1 | 9 | 3 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Eye injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 4 | 0 | 4 | 7 | 5 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Eschar (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 1 | 0
Procedural site reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 1
Transfusion-related circulatory overload (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 5
Periorbital haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Macroglossia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 2 | 2 | 3 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Atrial tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0
Nodal rhythm (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 2 | 0 | 2 | 3 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 2 | 2
Tachycardia (Cardiac disorders) | 3 | 0 | 0 | 2 | 1 | 1
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Coronary artery insufficiency (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ventricular hypokinesia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cranial nerve disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 9 | 1 | 1 | 11 | 4 | 0
Dizziness postural (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 3 | 0 | 3 | 4 | 3 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Facial paresis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 5 | 1 | 2 | 6 | 3 | 1
Memory impairment (Nervous system disorders) | 1 | 0 | 1 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 2 | 0 | 1 | 1 | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0 | 1 | 1 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Speech disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0
Tongue paralysis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Ageusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Akathisia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 1
Carotid artery thrombosis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Coordination abnormal (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nerve compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cerebellar syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypogeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1 | 2 | 0
Parkinson's disease (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Parkinsonism (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Partial seizures (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 6 | 0 | 2 | 13 | 5 | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | 0 | 2 | 2 | 3 | 0
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 9 | 2 | 1
Splenic lesion (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 12 | 2 | 6
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 9 | 2 | 4
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 1
Thymus disorder (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 2 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 3 | 1
Excessive cerumen production (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 1 | 0
External ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 1 | 0 | 0 | 0
Mastoid effusion (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 2 | 0 | 0 | 1 | 0 | 0
Eye disorder (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Retinal haemorrhage (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1
Retinal vascular disorder (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 3 | 1 | 0 | 1 | 0 | 0
Exophthalmos (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Blindness (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 5 | 0 | 0 | 0 | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 3 | 6 | 3 | 3
Abdominal rigidity (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 4 | 24 | 10 | 2
Diarrhoea (Gastrointestinal disorders) | 8 | 0 | 4 | 17 | 11 | 3
Dry mouth (Gastrointestinal disorders) | 3 | 1 | 2 | 5 | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 3 | 3 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 2 | 3 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0 | 1 | 3 | 2 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 1 | 4 | 24 | 14 | 5
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 1
Rectal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 4 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 3 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1 | 4 | 11 | 9 | 6
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Angina bullosa haemorrhagica (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 5 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Noninfective gingivitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oral mucosal blistering (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tongue haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Lip haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 2 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 2 | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 1 | 10 | 8 | 2 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 0 | 2 | 10 | 5 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0
Night sweat (Skin and subcutaneous tissue disorders) | 3 | 0 | 2 | 1 | 0 | 1
Onychomadesis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 6 | 1 | 2 | 3 | 5 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 0 | 4 | 12 | 5 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 3 | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 4 | 0 | 1 | 5 | 1 | 3
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 0 | 3 | 5 | 2 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 0 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 1 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 0 | 3 | 2 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nodular rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Prurigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Scab (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Skin erosion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Stasis dermatitis (Product Issues) | 0 | 0 | 0 | 0 | 1 | 0
Sticky skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Chronic papillomatous dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 2 | 3 | 3 | 0
Chromaturia (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 0 | 1 | 1 | 1 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 2 | 1 | 3 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 1 | 0 | 2 | 0 | 0 | 0
Urine odour abnormal (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 2 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 4 | 0 | 0
Urine flow decreased (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cushingoid (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 1 | 4 | 13 | 7 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 4 | 9 | 1 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 | 0 | 3 | 4 | 2 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 0 | 1 | 5 | 4 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 2 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 1 | 4 | 7 | 3 | 2
spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 0 | 0
Amyotrophy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Joint instability (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Bacterial vaginosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 4 | 0 | 1 | 0 | 0 | 1
Clostridium bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Furuncle (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Klebsiella bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Klebsiella infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Molluscum contagiosum (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 3 | 0 | 0 | 4 | 3 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Perineal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Phlebitis infective (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 0 | 1 | 3 | 0
Rash pustular (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 2 | 2 | 0 | 0
Skin infection (Infections and infestations) | 3 | 0 | 0 | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 3 | 2 | 0 | 2
Upper respiratory tract infection bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 1 | 4 | 3 | 2 | 1
Abscess oral (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Catheter site infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Corona virus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Cystitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0
Oral fungal infection (Infections and infestations) | 0 | 0 | 0 | 2 | 1 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 3 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Tinea infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection enterococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Lip infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 7 | 1 | 8 | 24 | 9 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 4 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 4 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 5 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 11 | 1 | 14 | 21 | 8 | 5
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0 | 1 | 13 | 0 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0 | 2 | 0 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 3 | 3 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 2 | 0 | 0 | 2 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0 | 9 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Note that the agreements are between the clinical sites and the Sponsor (or its agents), which restrict the clinical trial sites' rights to discuss or publish trial results after the trial is completed.

DOCUMENTS (2):
  • Study Protocol (2022-08-31): https://cdn.clinicaltrials.gov/large-docs/58/NCT02807558/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-09): https://cdn.clinicaltrials.gov/large-docs/58/NCT02807558/SAP_001.pdf